CLINICAL TRIAL: NCT02457208
Title: Studying the Blood Levels of First-line Anti-tuberculosis Drugs in Relation to Treatment Outcomes Among Newly Diagnosed Adults With Pulmonary Tuberculosis on the Thai-Myanmar Border
Brief Title: PK Study of Anti-TB Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMRU1407
Record Dates: First submitted 2015-04-22; First posted 2015-05-29 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Tuberculosis
Keywords: pharmacokinetics
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Protons; Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2HRZE/4HR (Experimental): 2HRZE/4HR
  * Intensive phase: 2 months HRZE - once daily
  * Continuation phase: 4 months HR - once daily
  Adults will be treated with fixed dose combination (FDC) tablets containing:
  Intensive phase (content per tablet)
  Isoniazid -75 mg,
  Rifampicin - 150 mg,
  Pyrazinamide - 400 mg,
  Ethambutol - 275 mg
  Continuation phase (content per tablet)
  Isoniazid 150 mg
  Rifampicin 300 mg
  *Drug dosing will be adjusted by patient body weight.
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)

INTERVENTIONS:
Drug: Isoniazid (H)
Drug: Rifampicin (R)
Drug: Pyrazinamide (Z)
Drug: Ethambutol (E)

SUMMARY:
This is a prospective descriptive and pharmacokinetic study will be conducted among newly diagnosed patients registered in the two SMRU TB clinics located on the Thai-Myanmar border. This study aims to recruit (1) 30 adults with HIV co-infection and (2) 30 adults without HIV co-infection in one year. Patients will be given the standard 6 month anti-TB drugs as per WHO guidelines.

DETAILED DESCRIPTION:
The threat of tuberculosis and HIV remains as major public health issues all over the world. Multi-drug resistant tuberculosis (MDR TB) is also a rising public health issue. Currently available standardized TB treatment is 6 months in duration. Previous pharmacokinetic and pharmacodynamic (PK/PD) studies of anti-TB drugs have shown that a number of factors such as HIV status, diabetes, malnutrition, age, sex, race, genetics (e.g. NAT2 polymorphisms), drug- drug interactions and food interactions may cause variation of the PK and/or the treatment outcome. But the findings are not persistent from one study to another, for example Chideya S. et al's study in Botswana showed that lower Cmax of anti-TB drugs frequently occurred in TB/HIV coinfected patients and low Cmax of pyrazinamide was related to poor treatment outcomes. On the other hand Requena-Méndez A. et al's study showed the variation of rifampin Cmax was not related to HIV. Large between-patient variability in PK parameters was recently shown to be strongly associated with TB treatment failures and possibly the emergence of drug resistant TB.

The primary objective of this study aims to describe the plasma drug levels of the first-line anti- tuberculosis drugs in two different pulmonary TB patient groups: (1) adults with HIV co-infection and (2) adults without HIV co-infection. The secondary objectives are to investigate the clinical, microbiological and immunological outcomes of the study participants in relation to the plasma drug level and to conduct full genome sequencing and spoligotyping of MTB strains.

Plasma drug levels from venous blood will be measured densely 13 times per day at two occasions: after the first dose on Day 1 and 6 weeks after treatment. Thereafter plasma drug levels will be measured at six hours post-dose on months 2, 3, 4, 5 and 6.

Clinical, microbiological and immunological parameters such as liver and renal function, CRP and LTA4G and sputum examination (smear microscopy, RNA PCR, culture) to monitor clinical progress will also be measured.

The analysis on the plasma drug level in relation to the clinical and microbiological outcomes will be carried out in order to describe the PK/PD of anti-TB drugs and clinical, microbiogical and immunological outcomes in consideration of any possible factors that would influence the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and microbiogical diagnosis of pulmonary TB
2. Males and females aged >18 years old
3. Willing to comply with study procedures including residing in the TB centre or nearby for six months
4. Written informed consent provided by participant

Exclusion Criteria:

1. TB treatment in the past
2. Known or suspected pregnancy
3. Enrolled for TB treatment at one of the study sites
4. Known hypersensitivity/intolerance to one or more of anti-TB drugs
5. The MTB strain that shown resistant to Rifampicin, which is the precursor marker of MDR TB detected by a MTB/Rif Xpert Assay
6. Biochemistry test result:

   1. Creatinine > 3 x upper limit of normal (ULN)
   2. bilirubin > 2.5 x ULN
   3. AST and/or ALT > 5 x ULN
7. Refuse to take HIV testing
8. The diagnosed TB patients who choose to take the treatment at a Thai hospital or a hospital in Myanmar
9. The proven non-TB patients by clinical and microbiological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Plasma drug levels of Rifampicin | 6 Months
  Rifampicin, Isoniazid, Pyrazinamide and Ethambutol in different study groups
Plasma drug levels of Isoniazid | 6 Months
Plasma drug levels of Pyrazinamide | 6 Months
Plasma drug levels of Ethambutol | 6 Month

SECONDARY OUTCOMES:
Time to negativity of M. tuberculosis | 6 Months
  Time to negativity of M. tuberculosis in relation to drug
Genotyping MTB strains | 6 Months
  Genotyping MTB strains in order to see any infection with new wild MTB or mutant strain in the study population

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand